CLINICAL TRIAL: NCT06359535
Title: An Economic Study on Prevention of Postoperative Nausea and Vomiting by HSK21542 Injection
Brief Title: An Economic Study of HSK21542 Injection for Prevention of Postoperative Nausea and Vomiting
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mengchang Yang (Other)
Responsible Party: Sponsor-Investigator, Mengchang Yang, Deputy Chief Physician, Sichuan Provincial People's Hospital
Organization: Sichuan Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSK21542-IIT-02
Record Dates: First submitted 2023-12-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSK21542-60μg (Experimental): HSK21542 injection of 60 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Interventions: Drug: HSK21542
- HSK21542-120μg (Experimental): HSK21542 injection of 120 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Interventions: Drug: HSK21542
- HSK21542-180μg (Experimental): HSK21542 injection of 180 μg was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Interventions: Drug: HSK21542
- Placebo (Placebo Comparator): A placebo was administered once within 15 min before the end of surgery, and was administered by intravenous bolus injection for no less than 30 s;
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK21542 — This study is an economic study and does not interfere with patients' medical treatment.
  Arms: HSK21542-120μg; HSK21542-180μg; HSK21542-60μg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study analyzed the efficacy and safety results of HSK21542 injection for the prevention of postoperative nausea and vomiting in a multicentre, randomized, double-blind, placebo-controlled dose-exploration study, as well as the real-world clinical routine use of troisisone and other (not limited to other setron drugs) for the prevention of postoperative nausea and vomiting and related adverse reaction treatment data. It was transformed into an effect indicator, and the possible costs involved in the study were analyzed, reasonable price parameters of HSK21542 injection were set, and the economic value of HSK21542 was explored.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old, male or female;
* The American Society of Anesthesiologists (ASA) Class I-III;
* 18 kg/m2 ≤ BMI ≤ 40 kg/m2;
* Hospitalized subjects scheduled to undergo elective laparoscopic abdominal or gynecological surgery under general anesthesia for an expected anesthetic time of ≥ 1 h;
* Subjects with intermediate or high risk (score ≥ 2 points) experiencing PONV judged by the investigator using the Apfel simplified risk score;
* Subjects who agree to participate in the trial and voluntarily sign the Informed Consent Form (ICF);

Exclusion Criteria:

* History or evidence of any of the following diseases prior to screening:Respiratory diseases: severe chronic obstructive pulmonary disease, acute exacerbation of chronic obstructive pulmonary disease, severe airway stenosis, large pharyngolaryngeal mass, (broncho) tracheoesophageal fistula or airway tear, and serious respiratory tract infection within 2 weeks prior to screening; Central nervous system disorders: subjects with epilepsy, Parkinson's disease, or other central nervous system diseases causing nausea and vomiting, such as craniocerebral injury, intracranial space-occupying lesions, intracranial aneurysms, etc.; Cardiovascular diseases: subjects with uncontrolled hypertension [systolic blood pressure (SBP) ≥170 mmHg and/or diastolic blood pressure (DBP) ≥105 mmHg without treatment with antihypertensive medication, or SBP ≥160 mmHg and/or DBP ≥100 mmHg after treatment with antihypertensive medications], serious cardiac insufficiency ( the New York Heart Association [NYHA] Grade III-IV), unstable angina pectoris, acute myocardial infarction, severe arrhythmia, history of tachycardia/bradycardia requiring medical treatment, Grade II-III atrioventricular block (excluding pacemaker use) within 6 months prior to screenin; Digestive disorders: subjects with intestinal obstruction or other digestive diseases that may cause nausea and vomiting as judged by the investigator; Patients with a confirmed diagnosis of vestibular function disorder, excluding travel sickness (including but not limited to peripheral vestibular syndrome, central vestibular syndrome, etc.); Subjects with a history of significant and chronic dizziness.
* Any of the following medications or treatments have been used at screening:Subjects who have received antiemetics/medications with antiemetic effects within 24 h before the start of surgery or who have used antiemetics/drugs with antiemetic effects before the start of surgery for no more than 5 half-lives (calculated as the longest time); Subjects with neoplasm malignant treated with chemotherapy within 4 weeks prior to screening;
* Laboratory test indicators at screening meet the following criteria:White blood cell count < 3.0 × 109/L;Platelet count < 80 × 109/L;Hemoglobin< 70 g/L;Prolongation of prothrombin time (PT) exceeding the upper limit of normal for 3 seconds;Prolongation of activated partial thromboplastin time (APTT) exceeding the upper limit of normal for 10 seconds;Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 3 × ULN;Total bilirubin > 2 × ULN;Blood creatinine > 2 × ULN;Fasting serum glucose≥ 11.1 mmol/L;
* Subjects anticipated to require continued endotracheal intubation after the end of surgery;
* Subjects anticipated to require the insertion of nasal or oral gastric tubes after the end of surgery;
* Subjects with a history of serious drug allergies or those allergic to the investigational drugs specified in the protocol;
* Subjects with a history of drug abuse, drug addiction, or alcoholism within 3 months prior to screening, where alcoholism is defined as consuming > 2 units of alcohol on average daily (1 unit = 360 mL of beer with 5% alcohol, 45 mL of liquor with 40% alcohol or 150 mL of wine);
* Subjects with nausea, retching, or vomiting within 24 h prior to induction of anesthesia (except for those caused by bowel preparation);
* Subjects who have participated in any investigational trial (defined as receiving investigational drug or placebo) within 3 months prior to screening;
* Female subjects who are pregnant or breastfeeding; female or male subjects of child-bearing potential are unwilling to use contraception throughout the entire study period and for 3 months after the study completion;
* Subjects judged by the investigator to be unsuitable for participating in this clinical trial for any other factors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2024-11-06 (Estimated); Study Completion 2024-11-06 (Estimated)

PRIMARY OUTCOMES:
Total direct medical costs, direct non-medical costs, indirect costs | 24 hours after the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mengchang Yang, Doctor, Principal Investigator — Prinipal Investigator
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Plan to publish articles to share data